CLINICAL TRIAL: NCT07328828
Title: Single-Center, Prospective, Single-Arm Clinical Study Protocol of Icaritin Soft Capsules as Adjuvant Therapy for Hepatocellular Carcinoma With High-Risk Recurrence Factors Post-Resection
Brief Title: Single-Arm Clinical Study of Icaritin Soft Capsules as Adjuvant Therapy for Hepatocellular Carcinoma Patients at High Risk of Postoperative Recurrence
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Collaborators: Hangzhou Zhongmei Huadong Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HCC-Icaritin-II-CN
Record Dates: First submitted 2025-06-19; First posted 2026-01-09 (Actual); Last update posted 2026-01-09 (Actual); Status verified 2025-06

CONDITIONS: RFS

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Study Cohort (Other): Within 8 weeks after R0 resection for hepatocellular carcinoma, patients begin adjuvant therapy with Icaritin Soft Capsules until disease recurrence, with treatment duration not exceeding 1 year. Icaritin Soft Capsules are administered orally at 600 mg twice daily, taken within 30 minutes after morning and evening meals with warm water. If a dose is missed and cannot be taken within 2 hours after a meal, patients should skip the missed dose and resume the next scheduled dose without make-up administration.
  Interventions: Drug: Icaritin soft capsules

INTERVENTIONS:
Drug: Icaritin soft capsules — Within 8 weeks after R0 resection for hepatocellular carcinoma, patients begin adjuvant therapy with Icaritin Soft Capsules until disease recurrence, with treatment duration not exceeding 1 year. Icaritin Soft Capsules are administered orally at 600 mg twice daily, taken within 30 minutes after morning and evening meals with warm water. If a dose is missed and cannot be taken within 2 hours after a meal, patients should skip the missed dose and resume the next scheduled dose without make-up administration.

SUMMARY:
Observing the Efficacy and Safety of Icaritin Soft Capsules as Postoperative Adjuvant Therapy in Hepatocellular Carcinoma Patients with High-Risk Factors for Recurrence (A Single-Arm, Single-Center, Prospective Clinical Study Protocol)

Detailed Description:

Primary Endpoint:

Recurrence-Free Survival (RFS)

Secondary Endpoints:

Recurrence-Free Survival Rate (RFSR) at 6 months and 12 months, Overall Survival (OS) , Quality of Life (QoL) , Safety (including incidence and severity of Adverse Events [AEs] and Serious Adverse Events [SAEs]).

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years.
* Clinically or histologically/cytologically confirmed hepatocellular carcinoma (HCC) per the Primary Liver Cancer Diagnosis and Treatment Guidelines (2022 Edition). Archived tissue samples are permitted; if no prior histological diagnosis exists, fresh tumor biopsy must be performed at baseline.
* At least one measurable lesion (RECIST v1.1).
* Child-Pugh score ≤ 7.
* Patients who underwent R0 resection (postoperative pathology report required) and showed no residual intrahepatic lesions on MRI within 8 weeks after surgery.
* At least one high-risk recurrence factor:
* Tumor size ≥ 5 cm;
* Tumor number ≥ 3;
* Microvascular invasion (MVI) grade: M1 or M2;
* Portal vein tumor thrombus resection (Cheng's classification I or II).
* No prior systemic therapy for HCC.
* Normal major organ function, with laboratory results meeting the following
* criteria within 7 days before treatment:
* Hemoglobin > 80 g/L;
* Absolute neutrophil count (ANC) ≥ 1.5 × 10⁹/L;
* Platelet count ≥ 40 × 10⁹/L;
* Serum albumin ≥ 28 g/L;
* Total bilirubin ≤ 2 × upper limit of normal (ULN);
* AST/ALT ≤ 5 × ULN;
* Alkaline phosphatase (ALP) ≤ 2.5 × ULN;
* Serum creatinine ≤ 1.5 × ULN and creatinine clearance ≥ 50 mL/min.
* Coagulation function: International normalized ratio (INR) ≤ 1.5 × ULN or prothrombin time (PT) ≤ 16 s.
* Ability to swallow and absorb oral medication.
* Negative serum pregnancy test within 7 days before randomization for women of childbearing potential; agreement to use effective contraception during treatment and for 60 days after the last dose.
* Voluntary participation with signed informed consent and expected good compliance.

Exclusion Criteria:

* Prior systemic therapy for HCC, including chemotherapy, targeted agents (e.g., sorafenib, lenvatinib, regorafenib), immune modulators (anti-PD-1/PD-L1/CTLA-4), or modern Chinese medicine with antitumor indications. Concurrent use of any investigational drug (except antiviral therapy) is excluded.
* Recurrent or metastatic HCC.
* Clinically significant ascites, pleural effusion, or pericardial effusion uncontrolled by medication at enrollment.

(Note: Imaging-detected ascites without clinical symptoms is permitted.)

* History of abdominal wall fistula, gastrointestinal perforation, refractory unhealed gastric ulcer, or active gastrointestinal bleeding within 6 months before enrollment.
* HCC lesion(s) ≥ 10 cm in any dimension (confirmed by BICR), > 10 lesions, or HCC volume ≥ 50% of liver volume; macrovascular portal vein tumor thrombosis.
* Major cardiovascular impairment within 12 months before treatment:
* NYHA Class II+ heart failure;
* Unstable angina, myocardial infarction, or stroke;
* Arrhythmia with hemodynamic instability;
* QTc interval > 480 ms.
* Any surgery within 28 days before the first dose.
* History or current diagnosis of coagulopathy, bleeding, or thrombotic disorders.
* Clinically significant liver disease, including active viral hepatitis, alcoholic hepatitis, decompensated cirrhosis, severe fatty liver, hereditary liver disease, liver atrophy, superior vena cava syndrome, or portal hypertension.

(Note: Portal hypertension without ascites, jaundice, or gastrointestinal bleeding may be considered.)

* Active autoimmune disease requiring systemic therapy within the past 2 years.
* Live vaccine administered within 30 days before the first dose.
* Hypersensitivity to any component of Epimedium Soft Capsules.
* Uncontrolled active HBV, HCV, or HDV infection; active tuberculosis.
* Pregnancy, lactation, or unwillingness to use contraception during the study.
* Any condition that may contraindicate the study drug, compromise data reliability, increase treatment risk, or affect compliance (e.g., metabolic disorders, abnormal lab results).
* Investigator judgement of unsuitability for the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2024-03-01 (Actual); Primary Completion 2025-03-01 (Actual); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
RFS | Follow-up will be conducted for up to 1 year, from baseline through study completion, with imaging assessments performed at protocol-defined intervals.
  For eligible subjects meeting all inclusion/exclusion criteria, study-related data collection will commence within 8 weeks after hepatocellular carcinoma resection. Enrolled patients will enter the treatment phase and receive Icaritin Soft Capsules as postoperative adjuvant therapy. Following treatment initiation, contrast-enhanced CT or MRI will be performed every 3 months (±7 days) to evaluate hepatic lesions and detect potential recurrence or metastasis.

CONTACTS AND LOCATIONS:
Locations (1):
- the Second Affiliated Hospital, Zhejiang University School of Medicine, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No